CLINICAL TRIAL: NCT06423742
Title: Consecutive Dual-Session tDCS in Chronic Subjective Severe to Catastrophic Tinnitus With Normal Hearing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongtan Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-11-009
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Tinnitus, Subjective
Keywords: Transcranial direct current stimulation; Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The participants were randomly allocated with three different arms (control, single-session, and dual session) using block to balance the size of each group. . Participants who assigned to the control group underwent dual sham stimulation per day, twice a week for 1 month. Patients were received sham and true stimulation once alternately in the single session group and two true stimulation per day in the dual session group for the same period as the control group. All subjects who enrolled this study were given a conventional treatment such as tinnitus retraining therapy, sound therapy using sound generator, and medications like clonazepam, selective serotonin reuptake inhibitors for patients who wanted to take for relief of symptoms.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Sham Comparator): The subjects in control group were received two consecutive sessions of sham stimulation twice a week for 4 weeks (8 sessions in total).
  Interventions: Device: Transcranial direct current stimulation
- single-session (Active Comparator): Patients enrolled to the single-session group received tDCS on one random session out of two consecutive sessions.
  Interventions: Device: Transcranial direct current stimulation
- dual-session (Experimental): In the dual-session group, the patients underwent two consecutives tDCS.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — The device used for tDCS in this study was DC-Stimulator Plus (NeuroConn GmbH, Ilmenau, Germany). The localization of stimulation area (DLPFC) was determined according to the 10/20 EEG system. Non-conducting, elastic head strap was placed around the head to prevent displacement during stimulation. The recording electrode covered with 5 x 7 cm sized traditional rectangular sponge was soaked with 6-7 mL of 0.9% NaCl saline solution per side and placed on the F3 (anode, left frontal) and F4 (cathode, right frontal) EEG location. Subjects were given 2 mA stimulation intensity for 20 min per session including fade-in and fade-out times for 20 seconds each. Interval between each session was 20 min. Sham procedure has been adopted a Fade In of current, Short Stimulation, Fade Out (FISSFO) protocol that consist of initial ramp up for 20 seconds, 2 mA stimulation for 40 seconds, and 20 seconds for ramp down. To check to impendence, brief current of 110 µA over 15ms every 550ms was delivered.

SUMMARY:
We aimed to analyze the effect of continuous dual session tDCS in patients with severe chronic subjective tinnitus without any evidence of hearing loss in terms of relief of tinnitus perception, distress, and loudness. Also, we investigated the difference in the maintenance duration of the tinnitus suppression effect of consecutive dual session tDCS compared to other groups followed up for 2 months.

DETAILED DESCRIPTION:
The participants were randomly allocated with three different arms (control, single-session, and dual session) using block to balance the size of each group. Pure tone audiometry, speech audiometry, tinnitogram (pitch matching, loudness, minimal masking level and residual inhibition), auditory evoked potential, THI, visual analogue scale (VAS) of loudness, awareness and annoyance, and BDI were evaluated as a baseline tests. Participants who assigned to the control group underwent dual sham stimulation per day, twice a week for 1 month. Patients were received sham and true stimulation once alternately in the single session group and two true stimulation per day in the dual session group for the same period as the control group. All subjects who enrolled this study were given a conventional treatment such as tinnitus retraining therapy, sound therapy using sound generator, and medications like clonazepam, selective serotonin reuptake inhibitors for patients who wanted to take for relief of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have experienced subjective tinnitus for over 3 months.
* Individuals with normal hearing, defined as an average pure tone threshold of less than 25 dB between 0.5-4 kHz, and the presence of the V wave at 30 dBnHL with a difference in V wave latency of less than 0.2 ms in both ears during the ABR test.
* Individuals with severe tinnitus, as indicated by a Tinnitus Handicap Inventory (THI) score of 58 or higher, and who have been assessed for symptoms of anxiety and depressive mood using the Beck Depression Inventory (BDI) questionnaire.

Exclusion Criteria:

* Those requiring treatment for neurological disorders such as epilepsy, migraine, or intracranial masses.
* Pregnant individuals on the day of providing consent and those with metal-based electric implantable prosthetics.
* Individuals with objective or somatic tinnitus, auditory hallucinations, unwillingness to provide written consent, or unwillingness to continue the trial, and those who have participated in previous trials involving tDCS for tinnitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) related to tinnitus | All participants were checked the VAS immediately after the last stimulation of every week for 4 weeks and 8th week (4 weeks after the end of treatment).
  To achieve a more quantitative evaluation of tinnitus reduction, we assessed the Visual Analog Scale (VAS).
Tinnitus Handicap Inventory (THI) | THI was assessed at the 4th and 8th week visits.
  The subjective improvement of tinnitus was evaluated using THI.
Beck depression inventory (BDI) | THI was assessed at the 4th and 8th week visits.
  To assess the association between tinnitus relief and depression, we evaluated the Beck Depression Inventory (BDI).

CONTACTS AND LOCATIONS:
Overall Officials: Sung Kyun Kim, Study Director — University of Michigan
Locations (1):
- Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do, South Korea